CLINICAL TRIAL: NCT07351604
Title: A Study on the Effectiveness of Large Language Model-Based Chatbot Interventions in Improving HPV Vaccine Awareness, Intention and Vaccination Rates
Brief Title: Effectiveness of Large Language Model-Based Chatbot in Improving HPV Vaccine Awareness, Intention and Vaccination Rates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Center for Disease Control and Prevention (Unknown)
Responsible Party: Principal Investigator, Jun Zhang, Professor, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HPV-AI-001
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: HPV Vaccination Rates; HPV Vaccine Awareness; HPV Vaccination Intention
Keywords: HPV vaccine; chatbot; Large language model; AI; HPV vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vaccine chatbot + Watching scientific videos group (Experimental): The chatbot will provide immediate, validated answers to participants' HPV vaccine-related questions. Scientific videos cover content related to HPV vaccine safety, efficacy, and other relevant information.
  Interventions: Device: Scientific videos; Device: Vaccine chatbot
- Watching scientific videos group (Experimental): Scientific videos cover content related to HPV vaccine safety, efficacy, and other relevant information.
  Interventions: Device: Scientific videos
- Vaccine chatbot group (Experimental): The chatbot will provide immediate, validated answers to participants' HPV vaccine-related questions.
  Interventions: Device: Vaccine chatbot
- Control group (No Intervention): No intervention

INTERVENTIONS:
Device: Scientific videos — Provide scientific videos related to HPV vaccine
  Arms: Vaccine chatbot + Watching scientific videos group; Watching scientific videos group
Device: Vaccine chatbot — Provide vaccine chatbot to answer HPV vaccine questions
  Arms: Vaccine chatbot + Watching scientific videos group; Vaccine chatbot group

SUMMARY:
This is an interventional study targeting parents of junior high school girls and female university students. The primary objective of the study is to evaluate the effectiveness of a vaccine chatbot in improving HPV vaccination rates. The secondary objectives are to evaluate the effectiveness in improving vaccine awareness and vaccination intention. All participants will be enrolled and randomly assigned to four groups: (1) vaccine chatbot plus scientific videos, (2) vaccine chatbot only, (3) scientific videos only, and (4) a control group (no intervention). The chatbot will provide immediate, validated answers to participants' HPV vaccine-related questions. The scientific videos will cover content related to HPV vaccine safety, efficacy, and other relevant information. The study will compare changes in HPV vaccine awareness, vaccination intention, and vaccination behavior between the intervention groups and the control group after the intervention to evaluate whether the three intervention strategies enhance HPV vaccine awareness, vaccination intention, and vaccination uptake.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of junior high school girls / Female university students.
2. Possess an electronic device with QR code scanning capability.
3. The daughters / female university students have no contraindications to HPV vaccination.
4. No mental disorders or visual/reading impairments; able to cooperate with and implement the corresponding intervention activities.
5. Have provided informed consent and are willing to participate in the study.

Exclusion Criteria:

-

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36000 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
HPV vaccination rates for eligible parents' daughters and female university students in all groups before and after the intervention | Baseline, two weeks and six months
  Whether participants' daughters and female university students get vaccinated against HPV or have an appointment for vaccination, measured by self-report and validated by vaccination information system

SECONDARY OUTCOMES:
HPV vaccine awareness for eligible parents' daughters and female university students in all groups before and after the intervention | Baseline and two weeks
  A questionnaire consisting of 11 questions related to HPV vaccines will be used to investigate the awareness of HPV vaccines.Total knowledge score is calculated based on the number of questions answered correctly by the participants and the higher scores mean a better outcome.
HPV vaccination intention for eligible parents' daughters and female university students in all groups before and after the intervention | Baseline and two weeks
  Parents' willingness to vaccinate their daughters against HPV and and female university students' willingness to vaccinate themselves, measured using a five-point Likert scale from "not willing at all" to "strongly willing"

OTHER OUTCOMES:
Vaccine chatbot acceptability and implementability | Two weeks
  A questionnaire consisting of 10 questions assessing usability and feasibility, fairness and safety, user experience, and overall assessment of the chatbot, measured using a five-point Likert scale from "not willing at all" to "strongly willing"
Factors influencing vaccination intention for eligible parents' daughters or female university students | Two weeks and six months
  Survey items: age, education level, marital status, occupation, annual income, and awareness of vaccines.